CLINICAL TRIAL: NCT03928067
Title: Online Intervention to Prevent Risky Behaviors During College Student Study Abroad Experiences
Brief Title: Brief Online Study Abroad Alcohol Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: RAND (Other)
Collaborators: Loyola Marymount University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01AA025909 (NIH)
Record Dates: First submitted 2019-04-22; First posted 2019-04-25 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Alcohol Abuse
Keywords: alcohol; sexual violence; risky sex; college students
MeSH Terms: conditions — Alcoholism | interventions — Syntex adjuvant formulation

STUDY DESIGN:
Masking Description: Masking of participants not possible
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TREK Study Abroad Program (Experimental): On-screen personalized normative feedback (PNF) will contain information on the drinking behavior and attitudes about gender- and country-specific study abroad peers. Participants will view text-based tips and strategies and watch clips of prior student abroad students discussing how they met their cultural engagement goals while abroad (Sojourner Adjustment Feedback or SAF). Content focuses around the four aspects of positive sojourner adjustment (social interaction with host nationals, cultural understanding and participation, language development and use, host culture identification) and the two negative sojourner adjustment factors while abroad (i.e., social interaction with co-nationals, homesickness/feeling out of place). The intervention will also contain text- and video-based tips and strategies for protective strategies used abroad to limit experience of risk sex and sexual violence victimization.
  Interventions: Behavioral: PNF + SAF
- Control (No Intervention): Control participants will receive a link to a general website offering study abroad advice (www.studyabroad.com) and will be asked to spend at least 20 to 30 minutes reviewing their institution's study abroad website content, including policies for drinking abroad. This control condition was selected as a form of "treatment as usual" as our conversations with study abroad personnel indicate this is the extent of typical information students receive about alcohol use abroad.

INTERVENTIONS:
Behavioral: PNF + SAF — Personalized normative feedback (PNF) to correct misperceived peer drinking norms abroad + sojourner adjustment feedback (SAF) to promote cultural engagement abroad.
  Other Names: TREK
  Arms: TREK Study Abroad Program

SUMMARY:
This study involves a randomized controlled trial that builds upon a successful pilot intervention study to address problematic and dangerous drinking among young adult college students studying abroad in foreign environments. Despite universities and colleges citing alcohol misuse as the most concerning issue for their students abroad, most institutions offer no empirically-based prevention efforts tailored to this at-risk population. The proposed intervention attempts to fill a major gap for the nearly 333,000 students completing study abroad programs each year by addressing empirically-based and theoretically-informed risk and protective factors of correcting misperceived peer drinking norms and promoting cultural engagement abroad. In addition to preventing heavy and problematic drinking, the intervention seeks to prevent risky behaviors and experience of sexual violence victimization, which are strikingly common among study abroad students and have the potential for lasting physical and psychological effects upon return home.

The investigators will conduct a randomized controlled trial of a developed intervention with a sample of 1,200 college students studying abroad from 35 U.S. universities and colleges. The brief, online intervention is text and video based and contains evidence-based components of personalized normative feedback to correct students' misperceived drinking norms, content to promote engagement with the cultural experience abroad and addressed difficulties adjusting to life in the foreign environment, and tips and strategies to prevent risky sexual behaviors and sexual violence victimization abroad. Participants will complete online surveys at five time points (predeparture, first month abroad, last month abroad, one-month post-return, and three-months post-return) to assess for intervention effects on drinking, risky sex, and sexual violence outcomes. The investigators will examine whether the mechanisms targeted by the intervention (changes in perceived norms, engagement in the cultural experience abroad) serve as mediators of intervention efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 25
* Signed up to study abroad in one of the 12 most popular destinations (i.e., United Kingdom, Italy, Spain, France, Germany, China, Ireland, Australia, Costa Rica, Japan, South Africa, and Mexico
* Plan to study abroad for between 8 and 21 weeks (approximately one quarter/semester)
* Have a working email address

Exclusion Criteria:

* None except not meeting eligibility criteria

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1200 (Estimated)
Dates: Start 2019-05-23 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Drinks per week | Past month (30 days)
  Total drinks per week in the past 30 days
Binge drinking frequency | Past month (30 days)
  Frequency of binge drinking (5+ drinks on one occasion for males; 4+ drinks on one occasion for females)
Alcohol-related consequences | Past month (30 days)
  24-item Brief Young Adult Alcohol Consequences Questionnaire, a measure of negative consequences often used with the college population. The scale contains 24 yes/no items that when summed gives a score from 0 to 24 (score of 24 indicates experience of all 24 alcohol consequences in the past 30 days)
Risky sexual behaviors | Past month (30 days)
  Sexual Risk Survey, a 23-item measure designed for and validated with college student samples. The scale yields an overall sexual risk behaviors score based on responses to the 23 items. The scale allows for open-ended responses that are then recoded into ordinal categories for generating an overall score from 0 to 92 (higher scores = higher risk).
Sexual violence victimization | Change in any sexual violence victimization experiences from before study abroad trip through the three months following the completion of the study abroad trip
  A scale to assess any sexual violence victimization was created from items modified and informed by items from the Sexual Experiences Survey and the National Drug-Facilitated, Incapacitated, and Forcible Rape study. The items are gender-specific (i.e., separate wording of items for those that identify as men, women, and gender-neutral) and contains 12 items with a yes/no format. Endorsement of any yes response yields an affirmative response to the outcome of experience of any sexual violence

CONTACTS AND LOCATIONS:
Locations (1):
- RAND, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pedersen ER, D'Amico EJ, LaBrie JW, Klein DJ, Farris C, Griffin BA. A randomized controlled trial of an online alcohol and sexual risk prevention program for college students studying abroad. J Subst Use Addict Treat. 2023 Feb;145:208951. doi: 10.1016/j.josat.2023.208951. Epub 2023 Jan 13. PMID 36880917
- [Derived] Pedersen ER, D'Amico EJ, LaBrie JW, Farris C, Klein DJ, Griffin BA. An online alcohol and risky sex prevention program for college students studying abroad: study protocol for a randomized controlled trial. Addict Sci Clin Pract. 2019 Aug 20;14(1):32. doi: 10.1186/s13722-019-0162-4. PMID 31429802